CLINICAL TRIAL: NCT02918175
Title: Technology to Improve Drug Adherence and Reinforce Guideline Based Exercise Targets in Patients With Heart Failure and Diabetes Mellitus (TARGET-HFDM)
Brief Title: Mobile Health Behavioral Intervention in Patients With Heart Failure and Diabetes Mellitus
Acronym: TARGET-HFDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00075572; 16SFRN30740010 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus; Heart Failure
Keywords: mHealth
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Intervention (Other): Subjects in this study arm will have data on activity levels, quality of life, medication adherence, and blood samples collected. In addition, they will receive personalized feedback on activity goals based on prior week step counts and participate in coaching sessions using the Pillbox medication tool.
  Interventions: Behavioral: mHealth
- No intervention (No Intervention): Subjects in this study arm will have data on activity levels, quality of life, medication adherence, and blood samples collected.

INTERVENTIONS:
Behavioral: mHealth — Personalized step count feedback and medication teaching tool.
  Other Names: Feedback on step counts; Duke PillBox medication adherence teaching tool
  Arms: mHealth Intervention

SUMMARY:
The overall objective of this study is to test a personalized mHealth intervention designed to increase physical activity and improve medication adherence in subjects with heart failure and diabetes mellitus. The study will leverage consumer technology as both an intervention and as a tool for data collection.

DETAILED DESCRIPTION:
This is a multi-center randomized controlled study in eligible subjects with heart failure and diabetes mellitus. Step counts, self-reported quality of life, medication adherence, blood samples and relevant clinical measures will be collected from all study subjects. The mobile health (mHealth) intervention will combine personalized text messages to encourage physical activity and a medication adherence teaching tool. A total of approximately 200 eligible subjects will be randomized in in a 1:1 ratio to either mHealth intervention + usual care/data collection or the control group (usual care/data collection only). The study duration is 6 months for all subjects; those in the intervention group will receive the mHealth intervention during the initial 3 months followed by 3 months of data collection only. The underlying hypotheses is that the proposed mHealth intervention can favorably impact specific health behaviors (physical activity and medication adherence) and physiologic measures of disease status for both heart failure and diabetes. Additional hypotheses to be tested will assess the persistence of behavioral changes (daily physical activity and medication adherence) and physiologic measures (NT-proBNP, HbA1c) beyond the 3-month time point of the active mHealth intervention (i.e. through 6 months).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Chronic heart failure, New York Heart Association (NYHA) class II-IV, with ongoing treatment with medications for heart failure for at least 1 month prior to enrollment
* Prior diabetes mellitus diagnosis, with ongoing treatment with anti-diabetes medications for at least 1 month prior to enrollment
* Adequate clinical stability in the judgment of the investigator to allow participation in study assessments and the intervention
* Independent with basic activities of daily living (ADLs), including the ability to ambulate independently
* No plan for revascularization (cardiac or peripheral), outpatient continuous intravenous inotrope administration, cardiac transplant or ventricular assist device implantation, or other cardiac surgery within 6 months of randomization
* Access to a compatible smart phone (iOS or Android)
* Signed informed consent

Exclusion Criteria:

* Acute myocardial infarction within prior 4 weeks
* Already actively participating in formal, facility-based cardiac rehabilitation
* Severe stenotic valvular disease (e.g., severe aortic stenosis)
* Implanted left ventricular assist device (LVAD)
* Recipient of a heart transplant
* Terminal illness other than heart failure with life expectancy < 6 months
* Impairment from stroke, injury or other medical disorder that precludes participation in the intervention
* Inability or unwillingness to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Change in mean weekly step count | from baseline to 3 months
  Increased activity

SECONDARY OUTCOMES:
Change in medication adherence score | from baseline to 3 and 6 months
  Improved medication adherence
Change in fill and refill performance rate | from baseline to 3 and 6 months
  Change in fill and refill performance rate
Change in mean weekly step count | from 3 to 6 months
  Increased activity
Change in NT-proBNP levels | from baseline to 3 to 6 months
  biomarkers
Change in HbA1C levels | from baseline to 3 to 6 months
  biomarkers
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | from baseline to 3 to 6 months
  QOL

OTHER OUTCOMES:
Change in plasma metabolic profile | from baseline to 3 months
  biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Felker, MD, Principal Investigator — Duke University Medical Center/Duke Clinical Research Institute
Locations (6):
- United States (6):
  - Stanford University School of Medicine, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Inova Health System, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No